CLINICAL TRIAL: NCT02194998
Title: Interferon-Free Therapy for Chronic Hepatitis C Virus Genotype 1 Infection in Participants With HIV-1 Coinfection Receiving Concurrent Antiretroviral Therapy (C_ASCENT)
Brief Title: Evaluating the Safety and Effectiveness of Interferon-Free Treatment of Hepatitis C Virus Infection in HIV-Coinfected Adults on Antiretroviral Therapy
Acronym: C_ASCENT
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study closed to accrual before the planned accrual goal was attained due to the availability of newer directly-acting antiviral (DAA) treatments for HCV.
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A5329; 11935 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 2014-07-17; First posted 2014-07-21 (Estimated); Results first posted 2019-06-04 (Actual); Last update posted 2021-11-04 (Actual); Status verified 2019-05

CONDITIONS: HIV Infections; Hepatitis C
MeSH Terms: conditions — HIV Infections; Hepatitis C | interventions — paritaprevir; dasabuvir; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Cohort A [INI-based ART + PTV/r/OBT + DSV +/- RBV 24 Weeks] (Experimental): Participants took an INI-based (RAL or DTG) ART regimen for HIV-1 and received the following medications for 24 weeks: paritaprevir/ritonavir/ombitasvir (PTV/r/OBT), dasabuvir (DSV), and ribavirin (RBV) (RBV for all participants (version 1) and only for participants with HCV genotype 1a (version 2)).
  Interventions: Drug: Paritaprevir/ritonavir/ombitasvir (PTV/r/OBT); Drug: Dasabuvir (DSV); Drug: Ribavirin (RBV)
- Cohort B [INI-based ART + PTV/r/OBT + DSV +/- RBV 12 Weeks] (Experimental): Participants took an INI-based (RAL or DTG) ART regimen for HIV-1 and received the following medications for 12 weeks: paritaprevir/ritonavir/ombitasvir (PTV/r/OBT), dasabuvir (DSV), and ribavirin (RBV) (RBV for all participants (version 1) and only for participants with HCV genotype 1a (version 2)).
  Interventions: Drug: Paritaprevir/ritonavir/ombitasvir (PTV/r/OBT); Drug: Dasabuvir (DSV); Drug: Ribavirin (RBV)
- Cohort C [PI-based ART + PTV/r/OBT + DSV +/- RBV 24 Weeks] (Experimental): Participants took a PI-based (DRV or ATV) ART regimen for HIV-1 and received the following medications for 24 weeks: paritaprevir/ritonavir/ombitasvir (PTV/r/OBT), dasabuvir (DSV), and ribavirin (RBV) (RBV for all participants (version 1) and only for participants with HCV genotype 1a (version 2)).
  Interventions: Drug: Paritaprevir/ritonavir/ombitasvir (PTV/r/OBT); Drug: Dasabuvir (DSV); Drug: Ribavirin (RBV)
- Cohort D [PI-based ART + PTV/r/OBT + DSV +/- RBV 12 Weeks] (Experimental): Participants took a PI-based (DRV or ATV) ART regimen for HIV-1 and received the following medications for 12 weeks: paritaprevir/ritonavir/ombitasvir (PTV/r/OBT), dasabuvir (DSV), and ribavirin (RBV) (RBV for all participants (version 1) and only for participants with HCV genotype 1a (version 2)).
  Interventions: Drug: Paritaprevir/ritonavir/ombitasvir (PTV/r/OBT); Drug: Dasabuvir (DSV); Drug: Ribavirin (RBV)

INTERVENTIONS:
Drug: Paritaprevir/ritonavir/ombitasvir (PTV/r/OBT) — PTV/r/OBT: 150/100/25 mg (two 75/50/12.5 mg fixed-dose combination tablets) orally once a day
Drug: Dasabuvir (DSV) — DSV: 250 mg orally twice a day
Drug: Ribavirin (RBV) — RBV: 1,000 or 1,200 mg (weight-based) dosed in two divided doses orally twice a day (all participants (version 1); only participants with HCV genotype 1a (version2))

SUMMARY:
HIV and hepatitis C virus (HCV) infection are diseases that share the same risk factors and routes of transmission. For this reason, many people infected with HIV are also infected with HCV. Interferon (IFN) is a drug used to treat HCV; however, in people coinfected with HIV and HCV, IFN treatment often does not work well and can cause unwanted side effects. The purpose of this study was to evaluate the safety, tolerability, and effectiveness of IFN-free HCV treatment in HIV/HCV coinfected adults who were taking antiretroviral (ARV) therapy.

DETAILED DESCRIPTION:
This study evaluated the safety, tolerability, and effectiveness of a combination of drugs to treat HCV in adults who were coinfected with HIV and HCV. The three drugs were paritaprevir/ritonavir/ombitasvir (PTV/r/OBT), dasabuvir (DSV), and ribavirin (RBV). In version 1 of the study, RBV was given to all participants. After revision in version 2, RBV was given only to participants with HCV genotype 1a; participants with HCV genotype 1b did not receive RBV.

This study enrolled HCV genotype 1a or 1b and HIV-1 coinfected participants (HCV treatment-naïve or HCV treatment-experienced) who were on a concurrent integrase inhibitor (INI)-based (raltegravir [RAL] or dolutegravir [DTG]) or protease inhibitor (PI)-based (darunavir [DRV] or atazanavir [ATV]) ART regimen. (The ART regimens were not provided by the study.) The participants were assigned to one of four cohorts (Cohorts A, B, C, and D). Participants in Cohorts A and B were on INI-based ART; participants in Cohorts C and D, on PI-based ART. For each group, the study proceeded in two steps: Step 1: on-HCV treatment and Step 2: post-HCV treatment follow-up. Participants in Cohorts A and C received the HCV drugs for 24 weeks; participants in Cohorts B and D, for 12 weeks. The target sample size goal was a total of 100 participants, with 25 participants per cohort.

Total study duration was up to 48 weeks. During Step 1 (on-HCV treatment), all participants had study visits at Weeks 2, 4, 6, 8, 10, and 12. Participants in Cohorts A and C had additional Step 1 study visits at Weeks 16, 20, and 24.

All participants had Step 2 (post-treatment follow-up) study visits 4, 12, and 24 weeks after registration to Step 2. Participants in Cohorts B and D had an additional Step 2 visit 36 weeks after registration to Step 2.

All study visits included a brief physical exam and blood collection. Select study visits included pregnancy testing for participants able to become pregnant, an electrocardiogram (EKG), an IFN gamma-induced protein 10 (IP-10) test, and collection of plasma samples.

Participants were able to coenroll in one of two optional substudies. In one substudy, participants attended two study visits at entry/Day 0 and Week 4 for 12-hour intensive pharmacokinetic (PK) sampling. In another substudy, participants underwent liver biopsies at two time points and PK sampling.

Study accrual was terminated early and participants who enrolled continued on study until completion.

ELIGIBILITY:
Inclusion Criteria:

* Men and women age greater than or equal to 18 to less than or equal to 70 years at study entry.
* Body mass index (BMI) from greater than or equal to 18 to less than 38 kg/m^2 within 42 days of study entry. BMI was calculated as weight measured in kilograms (kg) divided by the square of height measured in meters (m).
* HIV-1 infection
* CD4+ cell count greater than or equal to 200 cells/uL and CD4+ cell percentage greater than or equal to 14% within 42 days of study entry.
* On a stable, qualifying ART regimen for at least 8 weeks prior to entry.
* HIV-1 RNA less than 50 copies/mL for at least 6 months prior to study entry.
* Presence of chronic HCV infection defined as positive for anti-HCV antibody or HCV RNA at least 6 months before screening, and positive for HCV RNA at the time of screening; OR positive for HCV RNA at the time of screening with a liver biopsy consistent with chronic HCV infection any time prior to study entry.
* HCV treatment-naïve or unsuccessful treatment with pegylated or standard IFN alfa with or without RBV. NOTE: No prior exposure to HCV NS3/4A PI (including but not limited to TVR, BOC, simeprevir), NS5A inhibitors (including but not limited to daclatasvir or ledipasvir), NS5B NNI or NI inhibitors (including but not limited to sofosbuvir) was allowed.
* HCV genotype 1a or 1b infection
* Serum HCV RNA greater than 10,000 IU/mL obtained within 42 days prior to study entry.
* The following laboratory values obtained within 42 days prior to study entry.

  * Absolute neutrophil count (ANC) greater than or equal to 750/mm^3
  * Hemoglobin greater than or equal to 12 g/dL for men and greater than or equal to 11 g/dL for women
  * Platelet count greater than or equal to 90,000/mm^3
  * International normalized ratio (INR) less than or equal to 1.5
  * Participants with known inherited bleeding disorder and INR greater than or equal to 1.5 could be enrolled.
  * Calculated creatinine clearance (CrCl) using Cockcroft-Gault method greater than or equal to 60 mL/min
  * Alanine aminotransferase (ALT) less than or equal to 7 times the upper limit of the normal range (ULN)
  * Aspartate aminotransferase (AST) less than or equal to 7 times the ULN range
  * Total bilirubin less than 3 mg/dL for participants not on ATV and less than 6 mg/dL for participants on ATV
  * Direct bilirubin less than or equal to 1.5 times the ULN
  * Albumin greater than or equal to 3.5 g/dL
  * Serum alfa-fetoprotein (AFP) less than or equal to 100 ng/mL
* Classification of liver disease as cirrhotic or non-cirrhotic with no evidence of hepatocellular carcinoma according to specified criteria.
* For females of reproductive potential, a negative serum or urine pregnancy test with a sensitivity of less than or equal to 25 mIU/mL within 42 days prior to study entry.
* All participants must have agreed not to participate in a conception process (e.g., active attempt to become pregnant or to impregnate, sperm donation, in vitro fertilization).
* If participating in sexual activity that could lead to pregnancy, the participant (men and women) had to agree to use two reliable methods of contraception simultaneously.
* Participants who were not of reproductive potential were eligible without requiring the use of contraceptives.
* Ability and willingness of the participant to provide written informed consent.

Exclusion Criteria:

* Breastfeeding
* Pregnant sexual partner for male participants with HCV genotype 1a infection who would receive RBV. This criterion did not apply to male participants with HCV genotype 1b infection who would not receive RBV.
* Known allergy/sensitivity or any hypersensitivity to components of study drugs or their formulation.
* Acute or serious illness requiring systemic treatment and/or hospitalization within 42 days prior to study entry.
* Active hepatitis B infection (positive hepatitis B surface antigen [HBsAg]) within 42 days prior to study entry.
* History of decompensated liver disease (including but not limited to encephalopathy, variceal bleeding, or ascites) prior to study entry.
* Any cause of liver disease other than chronic HCV infection, including but not limited to the following: hemochromatosis, alpha-1 antitrypsin deficiency, Wilson's disease, autoimmune hepatitis, alcoholic liver disease, or drug-related liver disease.
* Uncontrolled or active depression or other psychiatric disorder within 24 weeks prior to study entry that in the opinion of the site investigator might preclude adherence to study requirements.
* Active drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements.
* Serious illness including uncontrolled seizure disorders, active coronary artery disease within 24 weeks prior to study entry, or other chronic medical conditions that in the opinion of the site investigator might preclude completion of the protocol.
* Presence of active or acute AIDS-defining opportunistic infections within 12 weeks prior to study entry.
* Active or history of malignancy within 5 years prior to study entry other than basal cell carcinoma of the skin and/or cutaneous Kaposi's sarcoma (KS) and/or cervical or anal dysplasia or carcinoma in situ.
* Clinically significant abnormal EKG, or EKG with QT interval corrected for heart rate (QTc) using Fridericia's correction formula (QTcF) greater than 450 msec within 42 days of study entry.
* Use of colony stimulating factors, such as granulocyte colony stimulating factor (GCSF) or erythropoietin within 42 days of study entry.
* Infection with any HCV genotype other than genotype 1, or mixed genotype infection any time prior to study entry.
* History of major organ transplantation with an existing functional graft any time prior to study entry.
* History of hemoglobinopathy (e.g., thalassemia) or any other cause of or tendency to hemolysis any time prior to study entry.
* Anticoagulants such as Coumadin (Warfarin), Dicumarol, Plavix (Clopidrogel), low-molecular weight Heparin, Lovenox (Enoxaparin), or Dabigatran (Pradaxa), aspirin, and Non-steroidal Anti-Inflammatory Drugs (NSAIDs) within 2 weeks prior to entry.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2015-09-16 (Actual); Primary Completion 2018-05-17 (Actual); Study Completion 2018-11-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark S. Sulkowski, MD, Study Chair — Johns Hopkins University
Locations (16):
- United States (15):
  - Alabama CRS, Birmingham, Alabama
  - UCLA CARE Center CRS, Los Angeles, California
  - University of Colorado Hospital CRS, Aurora, Colorado
  - Whitman-Walker Health CRS, Washington D.C., District of Columbia
  - Rush University CRS, Chicago, Illinois
  - Johns Hopkins University CRS, Baltimore, Maryland
  - New Jersey Medical School Clinical Research Center CRS, Newark, New Jersey
  - Weill Cornell Chelsea CRS, New York, New York
  - Cincinnati Clinical Research Site, Cincinnati, Ohio
  - Penn Therapeutics, CRS, Philadelphia, Pennsylvania
  - University of Pittsburgh CRS, Pittsburgh, Pennsylvania
  - The Miriam Hospital Clinical Research Site (TMH CRS) CRS, Providence, Rhode Island
  - Trinity Health and Wellness Center CRS, Dallas, Texas
  - Houston AIDS Research Team CRS, Houston, Texas
  - University of Washington AIDS CRS, Seattle, Washington
- Puerto Rico AIDS Clinical Trials Unit CRS, San Juan, Puerto Rico

REFERENCES:
- [Derived] Anthony DD, Sulkowski MS, Smeaton LM, Damjanovska S, Shive CL, Kowal CM, Cohen DE, Bhattacharya D, Alston-Smith BL, Balagopal A, Wyles DL. Hepatitis C Virus (HCV) Direct-Acting Antiviral Therapy in Persons With Human Immunodeficiency Virus-HCV Genotype 1 Coinfection Resulting in High Rate of Sustained Virologic Response and Variable in Normalization of Soluble Markers of Immune Activation. J Infect Dis. 2020 Sep 14;222(8):1334-1344. doi: 10.1093/infdis/jiaa254. PMID 32406487
- See also: DAIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table), Version 1.0, December 2004 (Clarification, August 2009). — http://rsc.niaid.nih.gov/sites/default/files/table-for-grading-severity-of-adult-pediatric-adverse-events.pdf
- See also: Manual for Expedited Reporting of Adverse Events to DAIDS (DAIDS EAE Manual), Version 2.0, January 2010. — http://rsc.niaid.nih.gov/sites/default/files/manual-exped-aes-v2_0.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from September 2015 to December 2016 at 16 U.S. sites.
Pre-assignment Details: There was no randomization in this study. Participants were stratified according to evidence of cirrhosis (yes versus no). The enrollment to the strata level for cirrhosis=yes was limited to no more than 30% within any particular study cohort.
Period: On-HCV Treatment
Arm/Group | Cohort A [INI-based ART + PTV/r/OBT + DSV +/- RBV 24 Weeks] | Cohort B [INI-based ART + PTV/r/OBT + DSV +/- RBV 12 Weeks] | Cohort C [PI-based ART + PTV/r/OBT + DSV +/- RBV 24 Weeks] | Cohort D [PI-based ART + PTV/r/OBT + DSV +/- RBV 12 Weeks]
Started | 21 | 6 | 15 | 4
Completed | 21 | 5 | 15 | 4
Not Completed | 0 | 1 | 0 | 0
Not completed — Did not pick up study medication | 0 | 1 | 0 | 0
Period: Post-HCV Treatment Follow-Up
Arm/Group | Cohort A [INI-based ART + PTV/r/OBT + DSV +/- RBV 24 Weeks] | Cohort B [INI-based ART + PTV/r/OBT + DSV +/- RBV 12 Weeks] | Cohort C [PI-based ART + PTV/r/OBT + DSV +/- RBV 24 Weeks] | Cohort D [PI-based ART + PTV/r/OBT + DSV +/- RBV 12 Weeks]
Started | 21 | 5 | 15 | 4
Completed | 20 | 5 | 14 | 4
Not Completed | 1 | 0 | 1 | 0
Not completed — Lost to Follow-up | 1 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Participants who initiated study treatment.
Groups:
- Cohort D [PI-based ART + PTV/r/OBT + DSV +/- RBV 12 Weeks]: Participants took a PI-based (DRV or ATV) ART regimen for HIV-1 and received the following medications for 12 weeks: paritaprevir/ritonavir/ombitasvir (PTV/r/OBT), dasabuvir (DSV), and ribavirin (RBV) (RBV for participants with HCV genotype 1a only; participants with HCV genotype 1b did not receive RBV).
- Total: Total of all reporting groups
Arm/Group | Cohort A [INI-based ART + PTV/r/OBT + DSV +/- RBV 24 Weeks] | Cohort B [INI-based ART + PTV/r/OBT + DSV +/- RBV 12 Weeks] | Cohort C [PI-based ART + PTV/r/OBT + DSV +/- RBV 24 Weeks] | Cohort D [PI-based ART + PTV/r/OBT + DSV +/- RBV 12 Weeks] | Total
Number analyzed (Participants) | 21 | 5 | 15 | 4 | 45
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 48 [40 to 49] | 50 [49 to 54] | 58 [55 to 61] | 55 [49 to 59] | 53 [47 to 58]
Age, Customized [Count of Participants; unit: Participants]
  30-39 years | 5 | 0 | 0 | 0 | 5
  40-49 years | 11 | 2 | 0 | 1 | 14
  50-59 years | 3 | 3 | 8 | 2 | 16
  60-69 years | 2 | 0 | 7 | 1 | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 1 | 3 | 2 | 13
  Male | 14 | 4 | 12 | 2 | 32
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White Non-Hispanic | 5 | 1 | 3 | 2 | 11
  Black Non-Hispanic | 6 | 3 | 8 | 1 | 18
  Hispanic (Regardless of Race) | 10 | 1 | 4 | 1 | 16
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 21 | 5 | 15 | 4 | 45
CD4 Count [Median (Inter-Quartile Range); unit: cells/mm^3] — Population: All participants who initiated treatment and had baseline CD4 result available.
  cells/mm^3
    number analyzed (Participants) | 20 | 5 | 15 | 4 | 44
    (all) | 752 [467 to 1064] | 674 [528 to 726] | 646 [466 to 849] | 525 [404 to 683] | 665 [464 to 894]
HIV-1 RNA [Count of Participants; unit: Participants]
  Greater than 40 copies/mL | 0 | 0 | 1 | 0 | 1
  Less than or equal to 40 copies/mL | 21 | 5 | 14 | 4 | 44
HCV RNA, continuous [Median (Inter-Quartile Range); unit: Log10 IU/mL] — Population: All participants who initiated treatment and had baseline HCV RNA result available.
  Log10 IU/mL
    number analyzed (Participants) | 21 | 5 | 14 | 4 | 44
    (all) | 6.5 [6.0 to 6.8] | 5.9 [5.1 to 6.3] | 6.5 [5.8 to 7.0] | 6.2 [5.9 to 6.5] | 6.4 [5.8 to 6.8]
HCV RNA, categorized [Count of Participants; unit: Participants] — Population: All participants who initiated treatment and had baseline HCV RNA result available.
  Participants
    number analyzed (Participants) | 21 | 5 | 14 | 4 | 44
    ≥6 million IU/mL | 6 | 1 | 6 | 0 | 13
    <6 million IU/mL | 15 | 4 | 8 | 4 | 31
HCV Genotype [Count of Participants; unit: Participants]
  1A | 16 | 5 | 13 | 4 | 38
  1B | 5 | 0 | 2 | 0 | 7
HCV Treatment Experience [Count of Participants; unit: Participants]
  Naive | 20 | 5 | 12 | 3 | 40
  Experienced | 1 | 0 | 3 | 1 | 5
Cirrhosis Status [Count of Participants; unit: Participants]
  Cirrhotic | 6 | 0 | 2 | 0 | 8
  Non-Cirrhotic | 15 | 5 | 13 | 4 | 37

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response at 12 Weeks After HCV Treatment Discontinuation (SVR12)
Description: SVR12 was defined as HCV RNA less than the assay LLOQ (<15 IU/mL) at 12 weeks post HCV treatment discontinuation.
  A two-sided 90% confidence interval was calculated for the percentage of participants with SVR12 response using Clopper-Pearson method.
  For those whose HCV early responses prior to SVR12 evaluation met the guidelines for HCV Virologic Failure (VF), their SVR12 outcome was defined as non-response. Those missing a HCV RNA result from the week 12 post HCV treatment discontinuation visit (and missing all subsequent evaluations) were considered non-responders. However, if HCV RNA evaluations subsequent to week 12 post treatment discontinuation were non-missing, then the first HCV RNA subsequent to week 12 post treatment discontinuation was instead used to define the primary outcome.
Time Frame: At 12 weeks after last dose of HCV study treatment. The duration for study treatment for Cohorts A and C and Cohorts B and D was 24 and 12 weeks, respectively.
Population: Participants who initiated study treatment.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A [INI-based ART + PTV/r/OBT + DSV +/- RBV 24 Weeks] | Cohort B [INI-based ART + PTV/r/OBT + DSV +/- RBV 12 Weeks] | Cohort C [PI-based ART + PTV/r/OBT + DSV +/- RBV 24 Weeks] | Cohort D [PI-based ART + PTV/r/OBT + DSV +/- RBV 12 Weeks]
Number analyzed (Participants) | 21 | 5 | 15 | 4
percentage of participants | 95.2 [79.3 to 99.8] | 60 [18.9 to 92.4] | 100 [81.9 to 100] | 100 [47.3 to 100]
Statistical Analysis 1: Comparison: Cohort A [INI-based ART + PTV/r/OBT + DSV +/- RBV 24 Weeks]; Null Hypothesis: Cohort A's SVR12 rate <= 70%; Test type: Superiority — A one-sided exact binomial test was used against a null rate of 70% at a significance level of 5%; p < 0.01, One-Sided Exact Binomial Test — No adjustments for multiple comparisons
Statistical Analysis 2: Comparison: Cohort B [INI-based ART + PTV/r/OBT + DSV +/- RBV 12 Weeks]; Null Hypothesis: Cohort B's SVR12 rate <= 70%; Test type: Superiority — A one-sided exact binomial test was used against a null rate of 70% at a significance level of 5%; p = 0.47, One-Sided Exact Binomial Test — No adjustments for multiple comparisons
Statistical Analysis 3: Comparison: Cohort C [PI-based ART + PTV/r/OBT + DSV +/- RBV 24 Weeks]; Null Hypothesis: Cohort C's SVR12 rate <= 70%; Test type: Superiority — A one-sided exact binomial test was used against a null rate of 70% at a significance level of 5%; p < 0.01, One-Sided Exact Binomial Test — No adjustments for multiple comparisons
Statistical Analysis 4: Comparison: Cohort D [PI-based ART + PTV/r/OBT + DSV +/- RBV 12 Weeks]; Null Hypothesis: Cohort D's SVR12 rate <= 70%; Test type: Superiority — A one-sided exact binomial test was used against a null rate of 70% at a significance level of 5%; p = 0.24, One-Sided Exact Binomial Test — No adjustments for multiple comparisons

2. Primary Outcome: Number of Participants With an Occurrence of Serious Adverse Events (SAEs) as Defined by International Conference on Harmonisation (ICH) Criteria
Description: Participants who experienced at least one observed SAEs as defined by ICH after initiating HCV study treatment through 30 days post date of last dose of HCV study treatment.
Time Frame: From treatment initiation to 30 days post date of last dose of HCV study treatment (whether planned or premature discontinuation). The duration for HCV study treatment for Cohorts A and C and Cohorts B and D was 24 and 12 weeks, respectively.
Population: Participants who initiated study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A [INI-based ART + PTV/r/OBT + DSV +/- RBV 24 Weeks] | Cohort B [INI-based ART + PTV/r/OBT + DSV +/- RBV 12 Weeks] | Cohort C [PI-based ART + PTV/r/OBT + DSV +/- RBV 24 Weeks] | Cohort D [PI-based ART + PTV/r/OBT + DSV +/- RBV 12 Weeks]
Number analyzed (Participants) | 21 | 5 | 15 | 4
Participants | 1 | 1 | 2 | 0

3. Primary Outcome: Number of Participants Who Prematurely Discontinued HCV Study Treatment for Any Reason Other Than HCV Virologic Failure (VF)
Description: HCV VF was defined as follows: confirmed increase from nadir in HCV RNA (defined as two consecutive HCV RNA measurements of >1 log10 IU/mL above nadir) at any time point; failure to achieve HCV RNA <LLOQ (<15 IU/mL) by week 6; confirmed HCV RNA ≥LLOQ (defined as two consecutive HCV RNA measurements ≥LLOQ (≥15 IU/mL)) at any point after HCV RNA <LLOQ during HCV treatment
Time Frame: From treatment initiation to either 24 weeks (for Cohort A and C) or 12 weeks (for Cohort B and D). The duration for HCV study treatment for Cohorts A and C and Cohorts B and D was 24 and 12 weeks, respectively.
Population: Participants who initiated study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A [INI-based ART + PTV/r/OBT + DSV +/- RBV 24 Weeks] | Cohort B [INI-based ART + PTV/r/OBT + DSV +/- RBV 12 Weeks] | Cohort C [PI-based ART + PTV/r/OBT + DSV +/- RBV 24 Weeks] | Cohort D [PI-based ART + PTV/r/OBT + DSV +/- RBV 12 Weeks]
Number analyzed (Participants) | 21 | 5 | 15 | 4
Participants | 1 | 1 | 0 | 0

4. Primary Outcome: Number of Participants With an Occurrence of Signs/Symptoms Grade 3 or Higher
Description: Participants with signs/symptoms of grade 3 or higher post treatment initiation.
  Participants with grade 3 sign/symptom prior to treatment initiation must have had one grade higher than pre-treatment to meet this outcome.
  Severity grading was based on DAIDS AE Grading Table, Version 1.0.
Time Frame: as for outcome 2
Population: Participants who initiated study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A [INI-based ART + PTV/r/OBT + DSV +/- RBV 24 Weeks] | Cohort B [INI-based ART + PTV/r/OBT + DSV +/- RBV 12 Weeks] | Cohort C [PI-based ART + PTV/r/OBT + DSV +/- RBV 24 Weeks] | Cohort D [PI-based ART + PTV/r/OBT + DSV +/- RBV 12 Weeks]
Number analyzed (Participants) | 21 | 5 | 15 | 4
Participants | 0 | 2 | 3 | 0

5. Primary Outcome: Number of Participants With an Occurrence of Diagnoses Leading to Premature HCV Study Treatment or HIV-1 Antiretroviral (ARV) Discontinuation.
Description: Participants who had diagnoses leading to premature HCV study treatment or HIV-1 ARV discontinuation post treatment initiation.
Time Frame: From treatment initiation to end of study follow-up at 48 weeks.The duration for HCV study treatment for Cohorts A and C and Cohorts B and D was 24 and 12 weeks, respectively. The duration for ARV treatment for all cohorts was 48 weeks.
Population: Participants who initiated study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A [INI-based ART + PTV/r/OBT + DSV +/- RBV 24 Weeks] | Cohort B [INI-based ART + PTV/r/OBT + DSV +/- RBV 12 Weeks] | Cohort C [PI-based ART + PTV/r/OBT + DSV +/- RBV 24 Weeks] | Cohort D [PI-based ART + PTV/r/OBT + DSV +/- RBV 12 Weeks]
Number analyzed (Participants) | 21 | 5 | 15 | 4
Participants | 0 | 1 | 0 | 0

6. Primary Outcome: Number of Participants With an Occurrence of Laboratory Abnormality Grade 3 or Higher.
Description: Participants with an observed laboratory abnormalities grade 3 or higher post treatment initiation.
  If entry (pre-treatment) lab result was grade 3, then a grade 4 result was required to meet this outcome.
  Severity grading was based on DAIDS AE Grading Table, Version 1.0.
Time Frame: as for outcome 2
Population: Participants who initiated study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A [INI-based ART + PTV/r/OBT + DSV +/- RBV 24 Weeks] | Cohort B [INI-based ART + PTV/r/OBT + DSV +/- RBV 12 Weeks] | Cohort C [PI-based ART + PTV/r/OBT + DSV +/- RBV 24 Weeks] | Cohort D [PI-based ART + PTV/r/OBT + DSV +/- RBV 12 Weeks]
Number analyzed (Participants) | 21 | 5 | 15 | 4
Participants | 5 | 3 | 3 | 0

7. Secondary Outcome: Number of Participants Who Experienced HIV-1 Virologic Failure (VF)
Description: HIV-1 VF was defined as two consecutive HIV-1 RNA results ≥ 200 copies/mL.
Time Frame: From treatment initiation to 4 weeks after last dose of HCV study treatment. HIV-1 RNA was measured at weeks 2, 4, 6, 8, 10, 12, 16, 20, 24, and 28. The durations for HCV study treatment for Cohorts A/C and Cohorts B/D were 24 and 12 weeks, respectively.
Population: Participants who initiated study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A [INI-based ART + PTV/r/OBT + DSV +/- RBV 24 Weeks] | Cohort B [INI-based ART + PTV/r/OBT + DSV +/- RBV 12 Weeks] | Cohort C [PI-based ART + PTV/r/OBT + DSV +/- RBV 24 Weeks] | Cohort D [PI-based ART + PTV/r/OBT + DSV +/- RBV 12 Weeks]
Number analyzed (Participants) | 21 | 5 | 15 | 4
Participants | 0 | 0 | 0 | 1

8. Secondary Outcome: Number of Participants With Selected HIV-1 Resistance Mutations Among Participants Who Experience HIV-1 Virologic Failure (VF)
Description: Participants with one or more genotype mutations in protease conferring major resistance to any HIV-1 Protease Inhibitors (PI) antiretroviral drug, from a plasma sample drawn following confirmed HIV-1 VF outcome.
Time Frame: At confirmation of HIV-1 virologic failure.
Population: Participants who experienced confirmed HIV-1 virologic failure (a single participant from Cohort D [PI-based + (3 DAA: 12 wks)]).
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A [INI-based ART + PTV/r/OBT + DSV +/- RBV 24 Weeks] | Cohort B [INI-based ART + PTV/r/OBT + DSV +/- RBV 12 Weeks] | Cohort C [PI-based ART + PTV/r/OBT + DSV +/- RBV 24 Weeks] | Cohort D [PI-based ART + PTV/r/OBT + DSV +/- RBV 12 Weeks]
Number analyzed (Participants) | 0 | 0 | 0 | 1
Participants | 0 | 0 | 0 | 0

9. Secondary Outcome: Levels of Soluble CD14 (sCD14)
Description: Levels of sCD14. Baseline was defined as the date of first treatment dose.
Time Frame: At baseline, end of HCV treatment (EOT), and 12 weeks post EOT. The EOT for Cohorts A and C and Cohorts B and D was 24 and 12 weeks, respectively.
Population: All participants who initiated treatment and had available data at the study visit.
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Cohort A [INI-based ART + PTV/r/OBT + DSV +/- RBV 24 Weeks] | Cohort B [INI-based ART + PTV/r/OBT + DSV +/- RBV 12 Weeks] | Cohort C [PI-based ART + PTV/r/OBT + DSV +/- RBV 24 Weeks] | Cohort D [PI-based ART + PTV/r/OBT + DSV +/- RBV 12 Weeks]
Number analyzed (Participants) | 21 | 4 | 15 | 4
ng/mL
  sCD14 at Baseline: number analyzed (Participants) | 21 | 4 | 14 | 4
  sCD14 at Baseline | 1,832.0 [1,401.5 to 2,401.9] | 2,226.8 [2,161.1 to 2,289.0] | 3,157.0 [2,293.4 to 4,135.1] | 3,092.0 [2,271.8 to 4,711.9]
  sCD14 at EOT: number analyzed (Participants) | 21 | 2 | 15 | 4
  sCD14 at EOT | 2,126.5 [1,663.4 to 4,029.7] | 1,132.8 [1,113.8 to 1,151.7] | 2,421.1 [1,862.2 to 4,362.0] | 2,801.3 [1,888.9 to 5,114.9]
  sCD14 at 12 weeks post EOT: number analyzed (Participants) | 19 | 3 | 14 | 4
  sCD14 at 12 weeks post EOT | 1,977.3 [1,374.8 to 3,458.1] | 1,367.4 [792.3 to 1,470.7] | 3,424.5 [1,765.8 to 3,908.0] | 2,608.3 [1,521.9 to 3,286.3]

10. Secondary Outcome: Change in Soluble CD14 (sCD14)
Description: Absolute change from baseline in sCD14 levels in plasma calculated as value at the later time point minus baseline value. Baseline was defined as the date of first treatment dose.
Time Frame: as for outcome 9
Population: All participants who initiated treatment and had available data at baseline and the respective post-baseline visit.
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Cohort A [INI-based ART + PTV/r/OBT + DSV +/- RBV 24 Weeks] | Cohort B [INI-based ART + PTV/r/OBT + DSV +/- RBV 12 Weeks] | Cohort C [PI-based ART + PTV/r/OBT + DSV +/- RBV 24 Weeks] | Cohort D [PI-based ART + PTV/r/OBT + DSV +/- RBV 12 Weeks]
Number analyzed (Participants) | 21 | 4 | 15 | 4
ng/mL
  Change from baseline to EOT: number analyzed (Participants) | 21 | 2 | 14 | 4
  Change from baseline to EOT | 307.6 [-190.4 to 1,752.6] | -1,063.2 [-1,147.8 to -978.6] | -380.3 [-1,488.0 to 887.8] | 318.2 [-2,003.7 to 2,023.7]
  Change from baseline to 12 weeks post EOT: number analyzed (Participants) | 19 | 3 | 13 | 4
  Change from baseline to 12 weeks post EOT | 145.2 [-173.6 to 526.7] | -894.2 [-1,524.2 to -659.6] | -22.6 [-593.8 to 828.5] | -987.0 [-1,691.8 to -483.7]

11. Secondary Outcome: Levels of IP-10 Concentration.
Description: Levels of IP-10 (Interferon gamma-induced protein 10) concentration in plasma. Baseline was defined as the date of first treatment dose.
Time Frame: as for outcome 9
Population: All participants who initiated treatment and had available data at the study visit.
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Cohort A [INI-based ART + PTV/r/OBT + DSV +/- RBV 24 Weeks] | Cohort B [INI-based ART + PTV/r/OBT + DSV +/- RBV 12 Weeks] | Cohort C [PI-based ART + PTV/r/OBT + DSV +/- RBV 24 Weeks] | Cohort D [PI-based ART + PTV/r/OBT + DSV +/- RBV 12 Weeks]
Number analyzed (Participants) | 21 | 4 | 15 | 4
pg/mL
  IP-10 at baseline: number analyzed (Participants) | 21 | 4 | 14 | 4
  IP-10 at baseline | 379 [172.7 to 537.8] | 120.2 [82.7 to 249.5] | 225.5 [119.9 to 628] | 196.4 [107.6 to 382.7]
  IP-10 at EOT: number analyzed (Participants) | 21 | 2 | 15 | 4
  IP-10 at EOT | 100.9 [62.8 to 184] | 60.4 [34.6 to 86.3] | 76.6 [52.2 to 124.2] | 182.6 [117.6 to 481.3]
  IP-10 at 12 weeks post EOT: number analyzed (Participants) | 18 | 3 | 14 | 4
  IP-10 at 12 weeks post EOT | 94.6 [68.3 to 190.2] | 85.5 [33 to 92.8] | 82.5 [71.9 to 142.1] | 159.5 [81.5 to 238.8]

12. Secondary Outcome: Change in IP-10 Concentration.
Description: Absolute change from baseline in IP-10 (Interferon gamma-induced protein 10) concentration in plasma, calculated as value at the later time point minus baseline value. Baseline was defined as the date of first treatment dose.
Time Frame: as for outcome 9
Population: All participants who initiated treatment and had available data at baseline and the respective post-baseline visit.
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Cohort A [INI-based ART + PTV/r/OBT + DSV +/- RBV 24 Weeks] | Cohort B [INI-based ART + PTV/r/OBT + DSV +/- RBV 12 Weeks] | Cohort C [PI-based ART + PTV/r/OBT + DSV +/- RBV 24 Weeks] | Cohort D [PI-based ART + PTV/r/OBT + DSV +/- RBV 12 Weeks]
Number analyzed (Participants) | 21 | 4 | 15 | 4
pg/mL
  Change from baseline to EOT: number analyzed (Participants) | 21 | 2 | 14 | 4
  Change from baseline to EOT | -244.4 [-333.1 to -87] | -22.2 [-32.2 to -12.2] | -116 [-201 to -49.4] | -61.1 [-263.5 to 372]
  Change from baseline to 12 weeks post EOT: number analyzed (Participants) | 18 | 3 | 13 | 4
  Change from baseline to 12 weeks post EOT | -127 [-301.9 to -55] | -29.1 [-32.9 to -13.9] | -83.1 [-184.5 to -53.3] | -114.9 [-261.7 to 91.6]

13. Secondary Outcome: Number of Participants With HCV Mutations Conferring Resistance to Any Component of the HCV Treatment Regimen
Description: Study team decided to remove this secondary outcome measure due to reduced interest in study treatment as a result of development and approval of newer DAA's.
Time Frame: From treatment initiation to 12 weeks post date of last dose of HCV study treatment. The duration for HCV study treatment for Cohorts A and C and Cohorts B and D was 24 and 12 weeks, respectively.
Population: No participants are included in this analysis. The outcome measure was withdrawn and no specimen testing was performed.
Arm/Group | Cohort A [INI-based ART + PTV/r/OBT + DSV +/- RBV 24 Weeks] | Cohort B [INI-based ART + PTV/r/OBT + DSV +/- RBV 12 Weeks] | Cohort C [PI-based ART + PTV/r/OBT + DSV +/- RBV 24 Weeks] | Cohort D [PI-based ART + PTV/r/OBT + DSV +/- RBV 12 Weeks]
Number analyzed (Participants) | 0 | 0 | 0 | 0

14. Secondary Outcome: Percentage of Participants With Sustained Virologic Response at 24 Weeks After HCV Treatment Discontinuation (SVR24)
Description: SVR24 was defined as HCV RNA less than the assay LLOQ (<15 IU/mL) at 24 weeks post treatment discontinuation.
  A two-sided 90% confidence interval was calculated for the percentage of SVR24 response using method of Clopper-Pearson.
  For those whose HCV early responses prior to SVR24 evaluation met the guidelines for HCV VF, their SVR24 outcome was defined as non-response. Those missing a HCV RNA result from the week 24 post HCV treatment discontinuation visit (and missing all subsequent evaluations) were considered non-responders. However, if HCV RNA evaluations subsequent to week 24 post treatment discontinuation were non-missing, then the first HCV RNA subsequent to week 24 post treatment discontinuation was instead used to define the primary outcome.
Time Frame: At 24 weeks after the date of last dose of HCV study treatment. The duration for study treatment for Cohorts A and C and Cohorts B and D was 24 and 12 weeks, respectively.
Population: Participants who initiated study treatment.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A [INI-based ART + PTV/r/OBT + DSV +/- RBV 24 Weeks] | Cohort B [INI-based ART + PTV/r/OBT + DSV +/- RBV 12 Weeks] | Cohort C [PI-based ART + PTV/r/OBT + DSV +/- RBV 24 Weeks] | Cohort D [PI-based ART + PTV/r/OBT + DSV +/- RBV 12 Weeks]
Number analyzed (Participants) | 21 | 5 | 15 | 4
percentage of participants | 90.5 [72.9 to 98.3] | 60 [18.9 to 92.4] | 93.3 [72.1 to 99.7] | 100 [47.3 to 100]
Statistical Analysis 1: Comparison: Cohort A [INI-based ART + PTV/r/OBT + DSV +/- RBV 24 Weeks]; Null Hypothesis: Cohort A's SVR24 rate <= 70%; Test type: Superiority — A one-sided exact binomial test was used against a null rate of 70% at a significance level of 5%; p < 0.01, One-Sided Exact Binomial Test — No adjustments for multiple comparisons
Statistical Analysis 2: Comparison: Cohort B [INI-based ART + PTV/r/OBT + DSV +/- RBV 12 Weeks]; Null Hypothesis: Cohort B's SVR24 rate <= 70%; Test type: Superiority — A one-sided exact binomial test was used against a null rate of 70% at a significance level of 5%; p = 0.47, One-Sided Exact Binomial Test — No adjustments for multiple comparisons
Statistical Analysis 3: Comparison: Cohort C [PI-based ART + PTV/r/OBT + DSV +/- RBV 24 Weeks]; Null Hypothesis: Cohort C's SVR24 rate <= 70%; Test type: Superiority — A one-sided exact binomial test was used against a null rate of 70% at a significance level of 5%; p < 0.01, One-Sided Exact Binomial Test — No adjustments for multiple comparisons
Statistical Analysis 4: Comparison: Cohort D [PI-based ART + PTV/r/OBT + DSV +/- RBV 12 Weeks]; Null Hypothesis: Cohort D's SVR24 rate <= 70%; Test type: Superiority — A one-sided exact binomial test was used against a null rate of 70% at a significance level of 5%; p = 0.24, One-Sided Exact Binomial Test — No adjustments for multiple comparisons

ADVERSE EVENTS:
Time Frame: From treatment initiation to off study at 48 weeks.
Description: At entry, all signs/symptoms and selected laboratory values were collected, regardless of grade. Post-entry, signs/symptoms of ≥ Grade 2 and ALT values of ≥ Grade 3 were collected. Signs/symptoms that lead to change in treatment, selected laboratory values, and events that lead to HIV or HCV treatment discontinuation or that meet expedited AE or ICH SAE guidelines were reported regardless of grade. The DAIDS AE Grading Table (V1.0) and Expedited AE Manual (V2.0) were used.
Arm/Group | Cohort A [INI-based ART + PTV/r/OBT + DSV +/- RBV 24 Weeks] | Cohort B [INI-based ART + PTV/r/OBT + DSV +/- RBV 12 Weeks] | Cohort C [PI-based ART + PTV/r/OBT + DSV +/- RBV 24 Weeks] | Cohort D [PI-based ART + PTV/r/OBT + DSV +/- RBV 12 Weeks]
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/5 | 0/15 | 0/4
Serious Adverse Events (participants affected / at risk) | 2/21 | 2/5 | 2/15 | 0/4
Other Adverse Events (participants affected / at risk) | 21/21 | 5/5 | 15/15 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A [INI-based ART + PTV/r/OBT + DSV +/- RBV 24 Weeks] (N=21) | Cohort B [INI-based ART + PTV/r/OBT + DSV +/- RBV 12 Weeks] (N=5) | Cohort C [PI-based ART + PTV/r/OBT + DSV +/- RBV 24 Weeks] (N=15) | Cohort D [PI-based ART + PTV/r/OBT + DSV +/- RBV 12 Weeks] (N=4)
Myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 0
Hemiparesis (Nervous system disorders) | 0 | 0 | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A [INI-based ART + PTV/r/OBT + DSV +/- RBV 24 Weeks] (N=21) | Cohort B [INI-based ART + PTV/r/OBT + DSV +/- RBV 12 Weeks] (N=5) | Cohort C [PI-based ART + PTV/r/OBT + DSV +/- RBV 24 Weeks] (N=15) | Cohort D [PI-based ART + PTV/r/OBT + DSV +/- RBV 12 Weeks] (N=4)
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 1 | 0
Eye pain (Eye disorders) | 0 | 0 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 5 | 0 | 2 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 1 | 0 | 1
Vomiting (Gastrointestinal disorders) | 3 | 1 | 1 | 0
Chest discomfort (General disorders) | 1 | 0 | 1 | 0
Chest pain (General disorders) | 1 | 0 | 2 | 1
Chills (General disorders) | 2 | 0 | 0 | 0
Fatigue (General disorders) | 7 | 1 | 2 | 1
Malaise (General disorders) | 3 | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 1 | 0 | 0
Pain (General disorders) | 1 | 1 | 0 | 0
Peripheral swelling (General disorders) | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 2 | 0 | 0 | 0
Secretion discharge (General disorders) | 0 | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 1 | 0 | 0
Latent syphilis (Infections and infestations) | 2 | 0 | 0 | 0
Otitis media acute (Infections and infestations) | 0 | 0 | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 11 | 2 | 4 | 0
Aspartate aminotransferase increased (Investigations) | 10 | 2 | 6 | 0
Blood alkaline phosphatase increased (Investigations) | 2 | 0 | 4 | 1
Blood bicarbonate decreased (Investigations) | 2 | 1 | 4 | 1
Blood bilirubin increased (Investigations) | 12 | 3 | 10 | 3
Blood creatinine increased (Investigations) | 3 | 0 | 4 | 1
Blood glucose decreased (Investigations) | 4 | 1 | 5 | 1
Blood glucose increased (Investigations) | 11 | 4 | 9 | 2
Blood potassium decreased (Investigations) | 2 | 1 | 2 | 1
Blood potassium increased (Investigations) | 2 | 1 | 0 | 0
Blood sodium decreased (Investigations) | 9 | 2 | 8 | 0
Blood uric acid increased (Investigations) | 9 | 2 | 5 | 0
Haemoglobin abnormal (Investigations) | 0 | 0 | 1 | 0
Haemoglobin decreased (Investigations) | 4 | 2 | 2 | 0
International normalised ratio increased (Investigations) | 1 | 0 | 1 | 0
Lipase increased (Investigations) | 9 | 1 | 4 | 0
Neutrophil count decreased (Investigations) | 3 | 0 | 2 | 1
Platelet count decreased (Investigations) | 4 | 0 | 2 | 0
Troponin I increased (Investigations) | 0 | 0 | 1 | 0
White blood cell count decreased (Investigations) | 1 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 1 | 3 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1 | 0
Burning sensation (Nervous system disorders) | 0 | 0 | 2 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 1 | 0
Headache (Nervous system disorders) | 3 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 2 | 0
Loss of consciousness (Nervous system disorders) | 0 | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 1 | 0
Bipolar disorder (Psychiatric disorders) | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1 | 0
Drug dependence (Psychiatric disorders) | 0 | 1 | 0 | 0
Nocturia (Renal and urinary disorders) | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 1 | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 3 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 0
Rash generalised (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In accordance with the Clinical Trials Agreement between NIAID (DAIDS) and company collaborators, NIAID (DAIDS) provides companies with a copy of any abstract, press release, or manuscript prior to submission for publication with sufficient time for company review and comment. The publication/other disclosure can be delayed for up to 30 additional business days for manuscripts and five (5) business days for abstracts, to preserve U.S. or foreign patent or other intellectual property rights

DOCUMENTS (2):
  • Study Protocol (2016-06-08): https://cdn.clinicaltrials.gov/large-docs/98/NCT02194998/Prot_001.pdf
  • Statistical Analysis Plan (2019-04-29): https://cdn.clinicaltrials.gov/large-docs/98/NCT02194998/SAP_000.pdf